CLINICAL TRIAL: NCT02493829
Title: A Phase I Study of B7.1 (CD80)/IL-2 Immune Gene Therapy for High Risk MDS RAEB-2 and Acute Myeloid Leukaemia Patients Unsuitable for Allogeneic Haematological Stem Cell Transplant
Brief Title: B7.1/IL-2 Leukaemia Cell Vaccine for Non-Transplant AML RFUSIN2-AML2 (NTX)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King's College London (Other)
Collaborators: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2494
Record Dates: First submitted 2015-06-09; First posted 2015-07-10 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Leukemia, Myeloid, Acute; Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AML Cell Vaccine (Experimental)
  Interventions: Biological: AML Cell Vaccine

INTERVENTIONS:
Biological: AML Cell Vaccine

SUMMARY:
The study will be an open label, single arm, phase I study intended to identify the safety and tolerability of "AML Cell Vaccine" given to eligible MDS RAEB-2 and AML patients who have achieved a best response of complete remission or partial remission following their first or second course of standard induction chemotherapy.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of MDS RAEB-2 or primary (de novo) or secondary AML defined according to the WHO classification either as a new diagnosis or as a relapse.
* Patients for whom the optimal therapy in CR1 would be to undergo allogeneic bone marrow transplantation, but for whom this procedure is either not recommended (e.g. due to comorbidities) or not available (e.g. lack of a suitable donor).

Key Exclusion Criteria:

* Patients with MDS RAEB-2 or AML and favourable prognostic profile (good risk cytogenetics: t(15;17)(q22;q12~21), inv16(p13q22)/t(16;16)(p13;q22), t(8;21)(q22;q22) or cytogenetically normal AML with NPM1 mutation and absence of Flt-3 ITD).
* Patients unsuitable for standard induction chemotherapy.
* Patients who have previously undergone or will be able to undergo allogeneic transplantation.
* Patients who have had previous or current treatment with any form of investigational immunotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-05 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Vaccine-related toxicity based on the NCI criteria V4.0 | 52 weeks
Frequency, severity of adverse events to the AML cell vaccine | 52 weeks